CLINICAL TRIAL: NCT04543175
Title: Taste Disorders and Their Relation to Body Mass Index, Food Frequency Questionnaire and Quality of Life in Breast Cancer Patients During Chemotherapy.
Brief Title: Taste Disorders and Their Relation to BMI, FFQ, and EORTC QLQ-BR23 in Breast Cancer Patients During Chemotherapy.
Status: Completed | Type: Observational
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Dr. Vanessa Fuchs Tarlovsky, Principal investigator, Hospital General de Mexico
Other Study IDs: DI/13/111/04/0249
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Taste Disorders; Dysgeusia; Ageusia; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Taste Disorders; Dysgeusia; Ageusia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chemotherapy breast cancer patients: Newly diagnosed breast cancer patients (clinical stages IA, IIA, IIB, IIIA and IIIB) before and after chemotherapy with the following drugs (Doxorubicin + Cyclophosphamide (DC) or Paclitaxel + Carboplatin (PC) or Docetaxel were followed until they complete four cycles of chemotherapy.
  Interventions: Other: Taste disorder´s test

INTERVENTIONS:
Other: Taste disorder´s test — Each patient performed their own test placing three drops with a disposable dropper from each bottle into the center of the tongue for whole-mouth testing.
  Other Names: Taste disorders

SUMMARY:
Taste disorders in cancer patients during chemotherapy could be consider as multifactorial disease, it is related with changes of food consumption. Approximately 36-69% of the patients under chemotherapy suffer oral toxicity or dysgeusia

A prospective case- only observational study was conducted in patients of the Hospital General de México for two years. A self-reported taste survey was used, and patients scored their results in a Likert scale.

ELIGIBILITY:
Inclusion Criteria:

- Chemotherapy with Doxorubicin + Cyclophosphamide (DC) or Paclitaxel + Carboplatin (PC) or Docetaxel.

Exclusión Criteria:

* No smokers Infections in oral cavity Acute respiratory diseases Gastro- oesophageal reflux disease Other types of cancer.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients of Oncology ward in Hospital General de Mexico between 20 and 60 years old with newly diagnosed breast cancer.
  and chemotherapy with Doxorubicin + Cyclophosphamide (DC) or Paclitaxel + Carboplatin (PC) or Docetaxel.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of taste disorders and perception of the four basic flavors | 21 days
  to assess the prevalence of taste alterations perception of the four basic flavors (sweet, salty, bitter and acidic) in newly diagnosed breast cancer patients (clinical stages IA, IIA, IIB, IIIA and IIIB) before and after chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de México, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No